CLINICAL TRIAL: NCT05594446
Title: Morphometric Study of the Legs and Feet of Diabetic Patients in Order to Collect Data Intended to be Used to Measure by Dynamometry the Pressures Exerted by Several Medical Compression Socks at the Level of the Forefoot
Status: Completed | Type: Observational
Sponsor: Sigvaris France (Industry)
Collaborators: Clin-Experts (Industry)
Responsible Party: Sponsor
Other Study IDs: 2022-A01136-37
Record Dates: First submitted 2022-10-16; First posted 2022-10-26 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Diabetes
Keywords: diabetes; compression stockings
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to collect morphometric data of legs and feet in diabetic patients in order to model in the laboratory the pressures exerted by compression stockings on different areas of the foot

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over the age of 18
* Patients with diabetes of any type, balanced or not, with or without a history of mal perforating
* Giving their oral agreement to participate after information

Exclusion Criteria:

* Patients seen in an emergency
* Patient with lower limb amputee (even partial)
* Patients with a foot wound, whatever the etiology of the wound
* Presence of lymphedema
* History of foot trauma with sequelae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The recruitment of participants will be done within the framework of the usual consultation of the participating doctor, among the population meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Collection of anthropometric measurements of the foot : Ankle circumference at thinnest point (cm) | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings
Collection of anthropometric measurements of the foot : Popliteal heel height (cm) | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings
Collection of anthropometric measurements of the foot : Circumference of the calf at the strongest point (cm) | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings
Collection of anthropometric measurements of the foot : Circumference of the forefoot at the level of the metatarsal heads (cm) | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings
Collection of anthropometric measurements of the foot : Radius of curvature estimated by a template, of the head of the first metatarsus (cm) | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings
Collection of anthropometric measurements of the foot : Radius of curvature estimated by a template, of the head of the last metatarsus (cm) | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings
Collection of anthropometric measurements of the foot : European shoe size | 3 minutes
  From the anthropometric data collected, measurements will be made on specific areas by a dynamometric method in the textile laboratory, in particular pressure measurements by different medical compression stockings. These pressure measurements will be estimates of the pressures exerted on areas at risk of the feet of diabetic patients by different medical compression stockings

CONTACTS AND LOCATIONS:
Overall Officials: Didier RASTEL, PhD, Principal Investigator — SELARL PHILANGIO
Locations (1):
- Rastel Didier, Grenoble, France

IPD SHARING:
Plan to Share IPD: No